CLINICAL TRIAL: NCT04888377
Title: Aspirin Supplementation for Pregnancy Indicated Risk Reduction in Nulliparas (ASPIRIN): Neurodevelopmental Follow-up Trial
Brief Title: ASPIRIN: Neurodevelopmental Follow-up Trial
Status: Completed | Type: Observational
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Thomas Jefferson University (Other); RTI International (Other); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: GN ASPIRIN Follow Up
Record Dates: First submitted 2021-04-28; First posted 2021-05-17 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-07

CONDITIONS: Neurodevelopmental Abnormality
Keywords: Pre-eclampsia; Low Dose Aspirin; ASPIRIN Trail; NICHD Global Network; Global Network; ASPRIN Follow Up; BSID-III; Family Resources and Context; ASQ-36; Neurodevelopmental delays; hypertensive disorders of pregnancy (HDP); Pre-term birth; LDA
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antenatal exposure to low dose aspirin: Mothers in the Global Networks ASPIRIN trial were given 81 mg of Aspirin throughout their pregnancy with the follow-up studies participant.
  Interventions: Drug: Aspirin
- Antenatal exposure to Placebo: Mothers in the Global Networks ASPIRIN trial were given placebo throughout their pregnancy with the follow-up studies participant.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Participant's mothers were administered 81mg of Aspirin throughout their pregnancy with the participant.
  Groups: Antenatal exposure to low dose aspirin
Drug: Placebo — Participant's mothers were administered placebo throughout their pregnancy with the participant.
  Groups: Antenatal exposure to Placebo

SUMMARY:
A total of 620 children will be enrolled in this study from six sites in sub-Saharan Africa, South Asia, and Latin America. Half of the children's mothers will have taken aspirin and half will have taken placebo. This will allow the researchers to compare results of the two groups of children and determine if children exposed antenatally to low dose aspirin will have scores on the Bayley Scales of Infant Development-III (BSID-III) examination at 36 months of life (+/-3months) that are not inferior to the child's peers who were not exposed (i.e., by no more than a margin of 4 points).

DETAILED DESCRIPTION:
An estimated 250 million children under the age of 511 worldwide are at risk for not achieving their developmental potential; 52.9 million children under five years of age in low- and middle-income country (LMIC) settings have neurodevelopmental delays. Compounding the issue is preterm birth (more common in LMICs) which has consistently been identified as a cause of neurodevelopmental delay. A recent review reported that out of the estimated 13 million preterm infants who survive beyond the first month, 0.9 million will suffer long term neurodevelopmental impairment, with 345,000 moderately or severely affected. This burden places a significant strain on the families, healthcare systems and societies that provide care for these children. Data from other Global Network participating sites (Guatemala, Democratic Republic of Congo, Zambia and Pakistan) also found strikingly high rates of stunting ranging from 44% to 66%, among infants and toddlers. Poverty additionally contributes to the attainment of optimal neurodevelopment. As such, any study of neurodevelopment should at least document these potential confounders.

Aspirin has been shown to predominantly affect both the COX-1 pathway which is involved in thrombosis and the COX-2 pathway, which affects inflammation through the production of Aspirin Triggered Lipoxins. More specifically, aspirin has been shown to inhibit the production of IL-6, IL-1B, CRP and TNF-α all of which have been shown to negatively affect child neurodevelopment and be involved in preeclampsia and preterm birth.

This will be a prospective masked matched cohort study of children between 33 and 39 months (mean 36 months) of age whose mothers were randomized in the ASPIRIN trial *NCT02409680* (1:1 Aspirin-Placebo), who will be evaluated using the BSID-III. Additionally, the Family Resources and Context questionnaire will be performed to adjust for the local context and the ASQ-3 will be administered as a secondary screen. Recognizing the significant role that preterm birth plays in neurodevelopment, the investigators will include 100 (50 in each group) children who were delivered before 37 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Mother was enrolled in the GN ASPIRIN trial
* Mother consented to be recontacted
* Child's parents or guardians are willing and able to give consent
* Child is between 33-39 months of age
* Child does not have significant congenital anomaly (blind or deaf) that would affect them from completing study assessments
* Child does not have other medical conditions that would preclude the child from completing study assessments.

Exclusion Criteria:

* The child does not meet the inclusion criteria.

Ages: 33 Months to 39 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of approximately 620 children, between 33 and 39 months of age, whose mothers were included in the ASPIRIN trial.
Sampling Method: Probability Sample
Enrollment: 666 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McClure, PhD, Principal Investigator — RTI International
Locations (14):
- United States (8):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Christiana Care, Newark, Delaware
  - Boston University, Boston, Massachusetts
  - Columbia University, New York, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - RTI International, Research Triangle Park, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- INCAP, Guatemala City, Guatemala
- India (2):
  - Jawaharlal Nehru Medical College, Belagavi
  - Lata Medical Research Foundation, Nagpur
- Aga Khan University, Karachi, Pakistan
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No
The plan is to release primary results from the study.

REFERENCES:
- [Derived] Hoffman MK, Goudar S, Dhaded S, Figueroa L, Mazariegos M, Krebs NF, Westcott J, Tikmani SS, Karim F, Saleem S, Goldenberg RL, Lokangaka A, Tshefu A, Bauserman M, Patel A, Das P, Hibberd P, Chomba E, Mwenchanya M, Carlo WA, Trotta M, Williams A, Moore J, Nolen T, Goco N, McClure EM, Lobo MA, Cunha AB, Derman RJ. Neurodevelopment of Children Whose Mothers Were Randomized to Low-Dose Aspirin During Pregnancy. Obstet Gynecol. 2024 Apr 1;143(4):554-561. doi: 10.1097/AOG.0000000000005514. Epub 2024 Jan 23. PMID 38262066

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin: Children of mothers who received 81mg low-dose aspirin daily beginning between 6 weeks 0 days and 13 weeks 6 days, until 37 weeks or delivery.
- Placebo: Children of mothers who received placebo daily beginning between 6 weeks 0 days and 13 weeks 6 days, until 37 weeks or delivery.
Period: Overall Study
Arm/Group | Aspirin | Placebo
Started | 343 | 323
Completed BSID-III Assessment | 330 | 312
Completed (Complete data for BSID-III Cognitive Composite Score) | 329 | 311
Not Completed | 14 | 12
Not completed — Incomplete Follow-up or No Study Data | 1 | 3
Not completed — Physician Decision | 6 | 6
Not completed — Withdrawal by Subject | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | Placebo | Total
Number analyzed (Participants) | 343 | 323 | 666
Age, Continuous [Mean (Standard Deviation); unit: months] — Age refers to the child at screening and is measured in months
  months | 37.5 (1) | 37.5 (0.9) | 37.5 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 155 | 328
  Male | 170 | 168 | 338
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 71 | 65 | 136
    Asian | 175 | 159 | 334
    Black or African American | 97 | 99 | 196
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 71 | 65 | 136
    Not Hispanic or Latino | 272 | 258 | 530
Maternal education [Count of Participants; unit: Participants] — Maternal education categories
  Participants
    No formal schooling | 52 | 44 | 96
    Years of schooling: 13 years or more | 34 | 41 | 75
    Years of schooling: 7-12 | 196 | 177 | 373
    Years of schooling: Less than 7 | 61 | 61 | 122

OUTCOME MEASURES:

1. Primary Outcome: Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Cognitive Composite Score
Description: Mean of the Bayley-III Cognitive Composite Score (standardized mean 100, SD 15, range 55-155) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 329 | 311
score on a scale | 96 (9.9) | 96.8 (10.4)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Assuming a non-inferiority margin of 4 points in the BSID-III cognitive score as clinically significant, and a true effect of LDA of not more than a 1 point decrease, a total sample size of 620 was determined to provide 80% power for a one-sided test for non-inferiority with a type I error of 5%. To test this secondary hypothesis, the sample size also provided over 90% power, at a two-sided type I error of 5%, to detect a difference of 4 points between LDA and placebo based on a two-sided test; Test type: Non-Inferiority — The primary hypothesis of non-inferiority was tested by calculating the mean difference between treatment arms and its associated 90% confidence interval for the primary outcome. If the lower bound of the 90% confidence interval was greater than -4, then LDA was assumed to be non-inferior to placebo. If non-inferiority were assumed, a one-sided t-test would test the benefit of LDA compared to placebo. All models controlled for site as the original randomization stratification factor; p = 0.25, ANCOVA — For each outcome, the adjusted mean difference between treatment groups and the associated 95% confidence interval based on an ANCOVA model is presented; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.2 to 0.6] — Mean difference is Aspirin-Placebo

2. Secondary Outcome: Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Cognitive Composite Score Less Than 70
Description: Number of participants with the Bayley-III Cognitive Composite score less than 70 (standardized mean 100, SD 15, range 55-155) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 329 | 311
Participants
  Participants with Score Greater than or Equal to 70 | 327 | 309
  Participants with Score Less than 70 | 2 | 2

3. Secondary Outcome: Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Cognitive Composite Score Less Than 1 Standard Deviation (SD) Below the Mean
Description: Number of participants with the Bayley-III Cognitive Composite score less than 1 SD below the sample mean (standardized mean 100, SD 15, range 55-155) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 329 | 311
Participants
  Participants with Scores Greater than or Equal to 1 Standard Deviation (SD) Below the Mean | 297 | 285
  Participants with Scores Less than 1 Standard Deviation (SD) Below the Mean | 32 | 26

4. Secondary Outcome: Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Language Composite Score
Description: Mean of the Bayley-III Language Composite Score (standardized mean 100, SD 15, range 45-155) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 328 | 306
score on a scale | 101.2 (13.2) | 100.4 (13.6)

5. Secondary Outcome: Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Language Composite Score Less Than 70
Description: Number of participants with the Bayley-III Language Composite score less than 70 (standardized mean 100, SD 15, range 45-155) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 328 | 306
Participants
  Participants with Score Greater than or Equal to 70 | 327 | 302
  Participants with Score Less than 70 | 1 | 4

6. Secondary Outcome: Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Language Composite Score Less Than 1 Standard Deviation (SD) Below the Mean
Description: Number of participants with the Bayley-III Language Composite score less than 1 SD below the sample mean (standardized mean 100, SD 15, range 45-155) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 328 | 306
Participants
  Participants with Scores Greater than or Equal to 1 Standard Deviation (SD) Below the Mean | 290 | 273
  Participants with Scores Less than 1 Standard Deviation (SD) Below the Mean | 38 | 33

7. Secondary Outcome: Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Motor Composite Score
Description: Mean of the Bayley-III Motor Composite Score (standardized mean 100, SD 15, range 45-155) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 326 | 308
score on a scale | 99.4 (13.2) | 100.1 (13.9)

8. Secondary Outcome: Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Motor Composite Score Less Than 70
Description: Number of participants with the Bayley-III Motor Composite score less than 70 (standardized mean 100, SD 15, range 45-155) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 326 | 308
Participants
  Participants with Score Greater than or Equal to 70 | 323 | 305
  Participants with Score Less than 70 | 3 | 3

9. Secondary Outcome: Bayley Scales of Infant and Toddler Development, 3rd Edition (Bayley-III) Motor Composite Score Less Than 1 Standard Deviation (SD) Below the Mean
Description: Number of participants with the Bayley-III Motor Composite score less than 1 SD below the sample mean (standardized mean 100, SD 15, range 45-155) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 326 | 308
Participants
  Participants with Scores Greater than or Equal to 1 Standard Deviation (SD) Below the Mean | 281 | 264
  Participants with Scores Less than 1 Standard Deviation (SD) Below the Mean | 45 | 44

10. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Communication Total Score
Description: Mean of the ASQ Communication Total Score (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
score on a scale | 52 (8.9) | 50.7 (10.2)

11. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Communication Total Score Less Than 1 Standard Deviation (SD) Below the Mean
Description: Number of participants with the ASQ Communication Total score less than 1 SD below the sample mean (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
Participants
  Participants with Scores Greater than or Equal to 1 Standard Deviation (SD) Below the Mean | 277 | 256
  Participants with Scores Less than 1 Standard Deviation (SD) Below the Mean | 53 | 58

12. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Gross Motor Total Score
Description: Mean of the ASQ Gross Motor Total Score (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
score on a scale | 47.8 (12) | 48.3 (12.6)

13. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Gross Motor Total Score Less Than 1 Standard Deviation (SD) Below the Mean
Description: Number of participants with the ASQ Gross Motor Total score less than 1 SD below the sample mean (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
Participants
  Participants with Scores Greater than or Equal to 1 Standard Deviation (SD) Below the Mean | 270 | 253
  Participants with Scores Less than 1 Standard Deviation (SD) Below the Mean | 60 | 61

14. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Fine Motor Total Score
Description: Mean of the ASQ Fine Motor Total Score (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
score on a scale | 39.6 (16.6) | 38.3 (16)

15. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Fine Motor Total Score Less Than 1 Standard Deviation (SD) Below the Mean
Description: Number of participants with the ASQ Fine Motor Total score less than 1 SD below the sample mean (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
Participants
  Participants with Scores Greater than or Equal to 1 Standard Deviation (SD) Below the Mean | 255 | 246
  Participants with Scores Less than 1 Standard Deviation (SD) Below the Mean | 75 | 68

16. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Problem Solving Total Score
Description: Mean of the ASQ Problem Solving Total Score (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
score on a scale | 40.2 (13.7) | 40.2 (13.7)

17. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Problem Solving Total Score Less Than 1 Standard Deviation (SD) Below the Mean
Description: Number of participants with the ASQ Problem Solving Total score less than 1 SD below the sample mean (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
Participants
  Participants with Scores Greater than or Equal to 1 Standard Deviation (SD) Below the Mean | 265 | 256
  Participants with Scores Less than 1 Standard Deviation (SD) Below the Mean | 65 | 58

18. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Personal Social Total Score
Description: Mean of the ASQ Personal Social Total Score (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
score on a scale | 45.5 (9.8) | 45.3 (10)

19. Secondary Outcome: Ages and Stages Questionnaire, 3rd Edition (ASQ-3) Personal Social Total Score Less Than 1 Standard Deviation (SD) Below the Mean
Description: Number of participants with the ASQ Personal Social Total score less than 1 SD below the sample mean (range 0-60) (lower scores indicating greater impairment)
Time Frame: At a single visit occurring between 33-39 months corrected age
Population: The analysis population includes all randomized infants with available data for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 330 | 314
Participants
  Participants with Scores Greater than or Equal to 1 Standard Deviation (SD) Below the Mean | 273 | 252
  Participants with Scores Less than 1 Standard Deviation (SD) Below the Mean | 57 | 62

ADVERSE EVENTS:
Time Frame: At a single visit occurring at 33-39 months corrected age
Arm/Group | Aspirin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/329 | 0/311
Serious Adverse Events (participants affected / at risk) | 0/329 | 0/311
Other Adverse Events (participants affected / at risk) | 0/329 | 0/311

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT04888377/Prot_SAP_000.pdf